

\*\*FOR CCI USE ONLY\*\*

Approved by the Beth Israel Deaconess Medical Center Committee on Clinical Investigations:

Consent Approval Date: 01/28/2019

Protocol Number: <u>2018P000044</u>



## INFORMED CONSENT FORM TO TAKE PART IN A RESEARCH STUDY

SUBJECT'S NAME:

TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after

Cardiac Surgery: A Pilot Study

PRINCIPAL INVESTIGATOR: Balachundhar Subramaniam, MD MPH

PROTOCOL NUMBER: 2018P000044

## INTRODUCTION:

- This is a research study;
- Your participation is voluntary;
- A research study includes only people who choose to take part;
- You may or may not benefit from participating in the study. However, your participation may help others in the future as a result of knowledge gained from the research;
- You may leave the study at any time;
- ➤ If you choose not to take part, or if you leave the study, your decision will in no way harm your relationship with any member of the research team or any other individuals at Beth Israel Deaconess Medical Center.

Please read this consent form carefully and ask the investigators or study staff to explain any words orinformation that you do not clearly understand. Once you read this consent form and understand what your participation in this study will involve, you will be asked to sign this form if you wish to take part. You will be given a signed copy of the form to keep for your records.

#### DISCLOSURE OF SPECIAL INTERESTS OF BIDMC AND INVESTIGATORS

This study is being conducted by Balachundhar Subramaniam, MD MPH. There is no external funding agency in this study. Neither BIDMC nor Dr. Subramaniam has any additional interests in this research project.

## WHOM TO CONTACT IF YOU HAVE QUESTIONS OR PROBLEMS

If you have any questions, concerns or complaints about this research or experience any problems, you should contact Dr. Balachundhar Subramaniam at [617] 754-2712.

## **PURPOSE**

Cardiac (heart) surgery is a procedure associated with moderate to severe pain after surgery. A big contributor to the overall pain is sternal pain, or pain on the chest at the site of the surgical incision.



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam. MD

MPH

PROTOCOL #: 2018P000044



Currently, pain after surgery is treated by pain-reducing medications called opioids that you receive through a vein in your arm. Administration of opioids may lead to a number of adverse events like nausea, vomiting, sedation, decreased bowel activity, and more severe complications such as issues with your lungs and breathing.

A regional analgesic block (an injection of pain medicine between the shoulder and rib muscles) has been shown to reduce pain after breast or chest trauma surgeries. The anesthetic bupivacaine (study medication) has been Food and Drug Administration (FDA) approved for blocks and is widely used. The efficacy of using an analgesic block to reduce pain and opioid use after cardiac surgery has not been studied in enough people yet.

In this study we want to determine whether use of a regional analgesic block with bupivacaine can help reduce the chest pain you may experience following heart surgery.

## STUDY PARTICIPANTS

You have been asked to be in the study because you are undergoing heart surgery. Approximately 80 patients will participate in this study at Beth Israel Deaconess Medical Center.

## **DESCRIPTION OF STUDY DETAILS**

If you agree to be in this study, you will be asked to read and sign this consent form. After you sign the consent form, the following things will happen:

- Screening Procedures: Screening procedures are tests and procedures that will be done to determine if you are eligible to take part in the research study. For this research study, the screening procedures include:
  - We will review of your medical records to ensure that you are appropriate to participate in the study and that you don't not have any sensitivities to the study medication.
- 2. <u>Randomization Procedures:</u> It is not clear at this time whether the medication used in this study would affect your pain after cardiac surgery. For this reason, the treatment plan offered to you will be picked by chance [like the flip of a coin]. You will not be able to choose which treatment you receive. The chances of receiving either of the treatments are approximately equal. After the randomization, you will be assigned to one of the following groups:
  - Group 1: Bupivacaine
  - Group 2: Placebo (Salt water)



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD MPH




Depending upon the group to which you are assigned, you may receive a placebo instead of the study medication. A placebo is an inactive saline solution that looks like the study drug, but a placebo contains no active medication. Placebos are used to help determine if the results of the study are truly from the study drug. Neither you nor your physician will know whether you will be receiving the study drug or the placebo. However this information can be learned in case of an emergency.

It is important to note that this study medication will be given *in addition to* the regular pain medications you might receive after cardiac surgery.

- 3. <u>Research Procedures</u>: If you qualify to take part in this research study, you will undergo these research procedures:
  - A) **Administration of the Study Medication**: As part of your participation, we will be administering the study medication at two different time periods: 1) shortly after your surgery when you are first in the intensive care unit, and 2) one day after your surgery. The study medication or placebo will be administered by a trained anesthesiologist.

At each time point you will be given a total of 20 cc or about two tablespoons of study medication injection on each side of your sternum (chest). Ultrasound will be used to guide the injection and confirm it is in the appropriate place between the shoulder and rib muscles.

- B) **Short Daily assessment**: We will ask you a few thinking and memory questions each day while you are in the hospital. This will take about 3-5 minutes.
- C) **Data Collection from your Medical Record**: We will be accessing your medical records in order to obtain information on how you are doing. Specifically we will be looking at the pain medications administered and your reported pain scores. This data is routinely collected by nurses as part of your stay in the hospital after surgery.

Other aspects of your surgery and care after surgery will occur as they normally would if you had decided not to participate in the study.

4. <u>Monitoring/Follow-Up Procedures</u>. Procedures performed to evaluate the effectiveness and safety of the research procedures are called "monitoring" or "follow-up" procedures. For this research study, the monitoring/follow-up procedures include:

We will monitor you for four days after surgery to see how you are doing. To do this we will review your medical records and speak with your doctors and nurses as necessary.



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD MPH


APPROVED BY THE

COMMITTEE ON CLINICAL INVESTIGATIONS
01/27/2020
APPROVAL EXPIRATION DATE

#### RISKS AND DISCOMFORTS

As a result of your participation in this study, you are at risk for side effects listed in this section. You should discuss these with the investigator and with your regular doctor if you choose.

Ultrasound is a very safe technology, and has no additional risks associated with it. The risks of bupivacaine include:

## More Common [>5% occurrence]

Constipation, nausea, vomiting

## <u>Less Common</u> [>1% but <5% occurrence]

- Abnormal nervous system function such as excitation, depression, numbness, tingling sensation, seizures, drowsiness, unconsciousness.
- Abnormal heart functions including abnormal rhythm, decreased heart rate, decreased blood pressure, or heart block

## Rare [<1% occurrence]

- Allergic reactions including hives, itching, redness, swelling, coughing, sneezing and breathing difficulty
- Persistent numbness, tingling and weakness at the site of administration

There is also a minor risk of hematoma (a bruise or collection of blood under the skin) associated with the administration of any block; however use of ultrasound to guide administration of the block lessens the possibility of this risk.

#### LOSS OF CONFIDENTIALITY

There is the potential for loss of confidentiality by participating in this study. Every effort will be made to protect the confidentiality of your identifiable information.

#### CONFIDENTIALITY

Information learned from your participation in this study and from your medical record may be reviewed and photocopied by the Food and Drug Administration (FDA) and/or other federal and state regulatory agencies, and the Committee on Clinical Investigations, the Human Subjects Protection Office and others involved in research administration of the Beth Israel Deaconess Medical Center with protection of confidentiality so far as permitted by applicable law. Information resulting from this study and from your medical record may be used for research purposes and may be published; however, you will not be identified by name in such publications.

#### **POSSIBLE BENEFITS**



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD MPH




It is not possible to predict whether you will benefit directly from participation in this study. However, your participation may help others in the future as a result of knowledge gained from the research.

## OTHER AVAILABLE OPTIONS

Taking part in this study is voluntary. Instead of being in this study, you can decide not to participate.

This research study is not meant to diagnose or treat medical problems. Participation in this research study does not take the place of routine physical examinations or visits to your regular doctor.

We recommend that you discuss these and other options with the investigator and your regular doctor so that you can make a well-informed decision about participating in this study.

## IF YOU DECIDE NOT TO TAKE PART IN THE STUDY

Participation in this study is voluntary. You have the right to decide not to take part in this study. If you choose to participate, you have the right to leave the study at any time. Your decision to not participate will not result in any penalties or loss of benefits to you. The investigators will tell you about new information that may affect your willingness to stay in this study.

If you decide not to participate in the study or decide to leave the study early, your decision will not affect your relationship with the research team or any other individual at Beth Israel Deaconess Medical Center.

#### INVESTIGATORS RIGHT TO STOP THE STUDY

The investigators have the right to end your participation in this study if they determine that you no longer qualify to take part, or if it would be dangerous for you to continue, or if you do not follow study procedures as directed by the investigators. Beth Israel Deaconess Medical Center or the funding source may stop the study at any time.

## **COSTS AND/OR PAYMENTS TO YOU**

## **COSTS COVERED BY STUDY**

You will not be charged for the drug Bupivacaine Hydrochloride, which is part of this research study. However, you and your insurance company will be charged for other tests, procedures or medications of this study that are considered standard treatment for your medical condition.

#### CO-PAYMENT/DEDUCTIBLE STATEMENT

You will be responsible for any co-payments or deductibles that are standard for your insurance coverage.



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD MPH




#### PAYMENTS TO YOU:

You will not be paid for your participation in this study.

## **COST OF RESEARCH RELATED INJURY:**

If you are injured as a direct result of your participation in this study you should contact the Investigator at the number provided under the section "Whom to Call if You Have Questions" in this form. You will be offered the necessary care to treat your injury. You or your insurance company will be billed for medical care and/or hospitalization related to this injury. You will be responsible for all co-payments and deductibles required under your insurance. BIDMC will consider reimbursement of injury related expenses not covered by your insurance on a case-by-case basis. At this time there is no plan to reimburse you for items such as lost wages or lost time from work. By signing this consent form you have not given up any legal rights.

## OTHER IMPORTANT INFORMATION

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a> as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# AUTHORIZATION FOR USE AND DISCLOSURE OF YOUR PROTECTED HEALTH INFORMATION

As part of this study, we will be collecting, using and sharing with others information about you. Please review this section carefully as it contains information about the federal privacy rules and the use and disclosure of your information.

## PROTECTED HEALTH INFORMATION [PHI]

By signing this informed consent document, you are allowing the investigators and other authorized personnel to use [internally at BIDMC] and disclose [to people and organizations outside the BIDMC workforce identified in this consent] health information about you. This may include information about you that already exists (for example: your medical records and other sources of health information, demographic information, the results of any laboratory tests, and mental health records (if applicable) as well as any new information generated as part of this study. This is your Protected Health Information.

PEOPLE/GROUPS AT BIDMC WHO WILL SHARE AND USE YOUR PROTECTED HEALTH INFORMATION

Your Protected Health Information may be shared with and used by investigators working on this study, including the supporting research team (such as research assistants and coordinators, statisticians, data managers, laboratory personnel, pharmacy personnel, and administrative assistants), and may also be shared and used by other health care providers at BIDMC who have treated you in the past and have information relevant to the research, or who provide services to you in connection with the research. Your Protected Health Information may also be shared with the



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD

**MPH** 




members and staff of the Committee on Clinical Investigations of Beth Israel Deaconess Medical Center, which is responsible for reviewing studies for the protection of the research subjects.

## PEOPLE/GROUPS OUTSIDE OF BIDMC WITH WHOM YOUR PROTECTED HEALTH INFORMATION WILL BE SHARED

We will take care to maintain confidentiality and privacy about you and your Protected Health Information. We may share your Protected Health Information with the following groups so that they may carry out their duties related to this study:

- Statisticians and other data monitors not affiliated with BIDMC
- Your health insurance company
- The Food and Drug Administration [FDA], the Department of Health and Human Services [DHHS], the National Institute of Health [NIH], the Office for Human Research Protections [OHRP], and other federal and state agencies that may have jurisdiction over the research
- Hospital and Clinical Research Accrediting Agencies

Those who receive your Protected Health Information during the course of the research may not be required by the federal privacy regulations to protect it, and they may make further disclosures to others and use your information without being subject to penalties under those laws.

## WHY WE ARE USING AND SHARING YOUR PROTECTED HEALTH INFORMATION

The main reason for using and sharing your Protected Health Information is to conduct and oversee the research as described in this Informed Consent Document. There are many other reasons beyond the research for which BIDMC may use or disclose your Protected Health Information. Not all of these reasons require your express written authorization. For example, we will use and share your Protected Health Information to ensure that the research meets legal, institutional and accreditation requirements and to conduct public health activities. The various ways in which BIDMC may use and disclose your protected health information without your authorization are explained in a document called the Notice of Privacy Practices. If you have not received a copy of BIDMC's Notice of Privacy Practices, please ask us for one and review it before signing this form. In addition to signing this document, you may also be asked to sign a BIDMC General Agreement form acknowledging that you have received the BIDMC Notice of Privacy Practices.

## No Expiration Date - Right to Withdraw Authorization

Your authorization for the use and disclosure of your Protected Health Information in this Study shall never expire. However, you may withdraw your authorization for the use and disclosure of your Protected Health Information at any time provided you notify the Principal Investigator in writing. If you would like to take back your authorization so that your Protected Health Information can no longer be used in this study, please send a letter notifying the Principal Investigator of your withdrawal of your authorization to <u>Dr. Balachundhar Subramaniam</u> at 330 Brookline Ave., Boston,



TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD MPH




MA 02215. Please be aware that the investigators in this study will not be required to destroy or retrieve any of your Protected Health Information that has already been used or disclosed before the Principal Investigator receives your letter, and they are permitted to continue to use and disclose your previously collected information as necessary to complete the research.

#### REFUSAL TO SIGN

Your clinical treatment may not be conditioned upon whether you sign the Authorization for Research. However, if you choose not to sign this informed consent document and authorization for the use and disclosure of your Protected Health Information, you will not be allowed to take part in the research study.

## RIGHT TO ACCESS AND COPY YOUR PHI

If you wish to review or copy your Protected Health Information as it is made part of your medical record, you may do so after the completion or termination of the study by sending a letter to the Principal Investigator requesting a copy of your Protected Health Information. You may not be allowed to inspect or copy your Protected Health Information until this study is completed or terminated.

## ADDITIONAL CONTACT FOR QUESTIONS OR CONCERNS

You may contact the Human Subjects Protection Office at [617] 975-8500 in the event that you would like to obtain information or to offer input about the research study. This office is independent of the investigator or investigator's research staff and can also assist with questions relating to your rights as a participant in research, which may include questions, concerns or complaints about your participation in the study.



| Medical Center |
|---|
| SUBJECT'S NAME: |
| TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for Postoperative Analgesia after Cardiac Surgery: A Pilot Study |
| PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD MPH |



# THE FOLLOWING PARAGRAPHS CONTAIN SOME STANDARD INFORMATION WHICH GENERALLY APPLIES TO INDIVIDUALS PARTICIPATING IN A RESEARCH STUDY.

## CONSENT FORM FOR CLINICAL RESEARCH

I have read the previous page[s] of the consent form and the investigator has explained the details of the study. I understand that I am free to ask additional questions.

If I wish additional information regarding this research and my rights as a research subject, or if I believe I have been harmed by this study, I may contact the Human Subjects Protection Office (HSPO).

I am aware that this is a research project and that unforeseen side effects may occur.

I understand that the Beth Israel Deaconess Medical Center has no formal program for compensating patients for medical injuries arising from this research. Medical treatment will be provided for injuries at the usual charge to me or to my insurer unless payment is otherwise provided for in this consent form.

I understand that participation in this study is voluntary and I may refuse to participate or may discontinue participation at any time without penalty, loss of benefits, or prejudice to the quality of care which I will receive.

| I acknowledge that no guarantees have been made to me regarding the results of the treatment inv this study, and I consent to participate in the study and have been given a copy of this form. | | | |
|---|---|---|---|
| Signature of Subject or<br>Legally Authorized Representative<br>(Parent if the subject is a minor) | Date | | |
| Relationship of Legally Authorized Represent | · | to ask questions | before signing, and |
| SIGNATURE OF IN | /ESTIGATOR/Co-Investigator | DATE | |
| PRINT INVESTI | GATOR'S/Co-Investigator's | NAME | _ |

A signing co-investigator must be listed on the study's approved Research Staffing Form at the time of consent.

Informed Consent – Part D CCI Form: 6-2017



| SUBJECT'S NAME: |
|-----------------------------------------------------------------|
| TITLE OF RESEARCH PROTOCOL: Pecto-Intercostal Fascial Block for |
| Postoperative Analgesia after Cardiac Surgery: A Pilot Study |
| PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD |
| MPH |
| PROTOCOL #: <b>2018P000044</b> |



## THE FOLLOWING SECTIONS ARE NOT NEEDED FOR ALL STUDIES AND SHOULD BE **UTILIZED AS INDICATED:**

| If the subject is able to speak and understand English but is not able to read or write |
|---|
| I was present during the entire oral presentation of the informed consent and witnessed the subject's agreement to participate in the study. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: ———— |
| If the subject is able to understand English but is not physically able to read or write or see |
| I was present during the entire oral presentation of the informed consent and witnessed the subject's agreement to participate in the study. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: |
| If the subject is not English speaking and signed the translated Short Form in lieu of the English consent document. |
| As someone who understands both English and the language spoken by the subject, I interpreted, in the subject's language, the researcher's presentation of the English consent form. The subject was given the opportunity to ask questions. |
| Signature of Interpreter: |
| Printed name of Interpreter: |
| Date: |